CLINICAL TRIAL: NCT04222920
Title: Adalimumab Dose Reduction Aiming Low Serum Concentration With Control of Disease Activity: a Single Blind, Non-inferiority, Randomised Clinical Trial
Brief Title: Adalimumab Dose Reduction Aiming Low Serum Concentration With Control of Disease Activity
Acronym: ADDORA-low
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Reade Rheumatology Research Institute (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADDORA-low
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Adalimumab; Rheumatoid arthritis; Therapeutic Drug Monitoring; Drug level; Dose reduction
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: Patients with rheumatoid arthritis treated with adalimumab for at least 28 weeks and a serum adalimumab concentration above 5 mg/L will be randomly assigned to dose reduction by extending their dosing interval aiming a drug level of 2 mg/L or aiming a drug level of 5 mg/L
Who Masked: Participant
Masking Description: The participants are kept ignorant of the group to which they have been assigned
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low serum drug concentration (Experimental): Adalimumab dose reduction aiming a drug level of 2 mg/L
  Interventions: Other: Dose reduction to 2mg/L; Drug: Adalimumab
- High serum drug concentration (Active Comparator): Adalimumab dose reduction aiming a drug level of 5 mg/L
  Interventions: Other: Dose reduction to 5mg/L; Drug: Adalimumab

INTERVENTIONS:
Other: Dose reduction to 2mg/L — Adalimumab dose reduction aiming drug concentration of 2mg/L
  Arms: Low serum drug concentration
Other: Dose reduction to 5mg/L — Adalimumab dose reduction aiming drug concentration of 5mg/L
  Arms: High serum drug concentration
Drug: Adalimumab — Adalimumab

SUMMARY:
Several prior studies have shown that dose reduction or discontinuation of tumor necrosis factor (TNF)-inhibitors, like adalimumab, is possible in substantial number of patients with a rheumatic disease without an increase in disease activity. Prior studies showed that patients with concentrations higher than 5 mg/L are overexposed to adalimumab and can safely reduce the dose. In the first phase of treatment, an adalimumab concentration of 5mg/L is needed to achieve adequate clinical response. However to control disease activity after 28 weeks, lower concentration than 5 mg/L are probably sufficient. Recent published data suggest that concentrations of 0.1-0.5 mg/L are enough to control TNF blockade in this state. Yet, a study which investigates the lowest effective drug serum concentration is missing so far. The hypothesis is that serum adalimumab concentration of 2 mg/L is sufficient to control disease activity.

DETAILED DESCRIPTION:
Biological agents are frequently prescribed to optimize rheumatoid arthritis care. In order to prevent joint destruction it is necessary to maintain remission or low disease activity. Up to now clinicians used to continue the initial treatment regimen to maintain remission or low disease activity. Since biologic therapy is expensive, and is associated with patient burden as dose dependant risk for serious infections, multiple studies have been performed to show that a large proportion of patients with rheumatoid arthritis with stable low disease activity can reduce their dose without relapse of disease. In addition the latest European and American recommendations pose to reduce the dosage or to discontinue the bDMARDs in case of persistent remission or low disease activity. Yet, there are no recommendations on how this should be carried out.

Currently, most clinicians use Disease Activity Score in 28 joints (DAS28) and the Clinical Disease Activity Index (CDAI) to monitor dose reduction strategies. Although disease activity guided dose reduction is safe and cost-effective, a relatively novel strategy is dose reduction using serum drug concentrations (therapeutic drug monitoring). Most biologics are characterized by wide variation in pharmacokinetics between patients, resulting in wide range of drug concentrations when administered at the labeled dose. Therapeutic drug monitoring can be a valuable tool for optimizing the dosage of biopharmaceuticals and improving patient care on individual level. In other autoimmune diseases, such as inflammatory bowel disease, it is thought to be superior to empirical dose reduction and is already applied in clinical practice.

The rationale behind therapeutic drug monitoring is that medication dose correlates with serum drug levels and drug concentration correlates with therapeutic effect. The latter notion is demonstrated for adalimumb by Pouw et al. Adalimumab serum concentration in a range 5-8 mg/L is sufficient for adequate response. In the first phase of treatment, drug concentration must be high enough to control immunogenicity. To control disease activity in the 2nd phase (after 28 weeks), lower concentrations than 5 mg/L are probably sufficient. Our study group illustrated in 2018 that reducing adalimumab dose by prolonging the dosing interval with 50%, is non-inferior to continuation in patients with adalimumab levels > 8mg/L. In addition, recent published data suggest that concentrations of 0.1-0.5 mg/L are enough to control TNF in this phase. Since around 70% of the patients have adalimumab concentration above 5 mg/l, while an adalimumab concentration of 5 mg/L is enough for adequate response (7), a large extent of patients might thus be overexposed.

The hypothesis is that 1/ tapering adalimumab in RA patient doing well after 28 weeks using TDM aiming at 5mg/l (and disease activity measurement) results in maintenance of disease control and lower adalimumab use, and that 2/ tapering to a lower target drug level of 2 mg/L is non inferior to the higher 5mg/l target with respect to disease activity control and safety, and superior in adalimumab reduction. Tapering to achieve these lower targets (for example direct doubling of interval in patients with levels > 10 mg/L) might result in the lowest effective drug dose.

Disease activity after dose reduction, aiming adalimumab concentration of 2 mg/L or 5 mg/L, in rheumatoid arthritis patients treated with adalimumab for at least 28 weeks and a serum adalimumab concentration above 5 mg/L, will be evaluated in this multi-centre, randomized, single blinded trail. Patients with an adalimumab concentration above 5mg/L will be randomly assigned to dose reduction by extending their dosing interval aiming a drug level of 2 mg/L or aiming a drug level of 5 mg/L. A newly developed algorithm is used to determine the interval prolongation for each patient

Data regarding disease status, functioning, adalimumab serum concentrations, anti-drug antibodies and medical costs will be collected during this study.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis patient, according to ACR 1987 or ACR/EULAR 2010
* Treated for at least 28 weeks with adalimumab
* Adalimumab trough concentration >5mg/L
* Who has agreed to participate (written informed consent);
* Age 18 years or older.

Exclusion Criteria:

* scheduled surgery during the follow-up of the study or other pre-planned reasons for treatment discontinuation
* life expectancy shorter than follow-up period of the study;
* other disease that might flare if adalimumab is tapered like psoriasis, inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Mean time weighted DAS28-CRP | after 24 weeks
  The difference in mean time weighted DAS28-CRP after 28 weeks between dose reduction aiming serum adalimumab concentration of 5mg/L and 2mg/L

SECONDARY OUTCOMES:
Mean time weighted DAS28-CRP | after 12 weeks
  The difference in mean time weighted DAS28-CRP after 28 weeks between dose reduction aiming serum adalimumab concentration of 5mg/L and 2mg/L
Number of flares | after 24 weeks
  Cumulative incidence of flare is calculated in both groups
Direct medical costs | after 24 weeks
  Direct medical costs (medication, visits, cost TDM testing) at the separate time points
Drug levels | after 12 and 24 weeks
  The difference in drug levels between the measured drug level and the predicted drug level with the (newly developed) algorithm at different timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Gertjan Wolbink, MD, PhD, Principal Investigator — Reade Rheumatology Research Institute
Locations (1):
- Reade Rheumatology Research Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
To avoid duplication of research, the gathered data will be shared once all desirable data analysis have been performed and the results are published
Supporting Information: Study Protocol, SAP
Time Frame: Six months after the study is published the data will be shared
Access Criteria: Researchers with demonstrable interest in autoimmunity, biologicals, or TDM can contact the investigators of the trial if they are interested in gaining access to the data. Depending on their research objectives the data will be shared

REFERENCES:
- [Background] Chen DY, Chen YM, Hsieh TY, Hung WT, Hsieh CW, Chen HH, Tang KT, Lan JL. Drug trough levels predict therapeutic responses to dose reduction of adalimumab for rheumatoid arthritis patients during 24 weeks of follow-up. Rheumatology (Oxford). 2016 Jan;55(1):143-8. doi: 10.1093/rheumatology/kev298. Epub 2015 Aug 31. PMID 26324949
- [Background] Kievit W, van Herwaarden N, van den Hoogen FH, van Vollenhoven RF, Bijlsma JW, van den Bemt BJ, van der Maas A, den Broeder AA. Disease activity-guided dose optimisation of adalimumab and etanercept is a cost-effective strategy compared with non-tapering tight control rheumatoid arthritis care: analyses of the DRESS study. Ann Rheum Dis. 2016 Nov;75(11):1939-1944. doi: 10.1136/annrheumdis-2015-208317. Epub 2016 Jan 13. PMID 26764260
- [Background] l'Ami MJ, Krieckaert CL, Nurmohamed MT, van Vollenhoven RF, Rispens T, Boers M, Wolbink GJ. Successful reduction of overexposure in patients with rheumatoid arthritis with high serum adalimumab concentrations: an open-label, non-inferiority, randomised clinical trial. Ann Rheum Dis. 2018 Apr;77(4):484-487. doi: 10.1136/annrheumdis-2017-211781. Epub 2017 Sep 22. PMID 28939629
- [Background] Pouw MF, Krieckaert CL, Nurmohamed MT, van der Kleij D, Aarden L, Rispens T, Wolbink G. Key findings towards optimising adalimumab treatment: the concentration-effect curve. Ann Rheum Dis. 2015 Mar;74(3):513-8. doi: 10.1136/annrheumdis-2013-204172. Epub 2013 Dec 10. PMID 24326008